CLINICAL TRIAL: NCT05663801
Title: Efficacy Of Magnesium Sulphate Versus Ketamine as an Adjuvant to Bupivacaine in Pectoral Nerve Block During Mastectomy : Comparative Controlled , Randomized Double-Blind Study
Brief Title: Magnesium Sulphate Versus Ketamine as an Adjuvant to Bupivacaine in Pectoral Nerve Block During Mastectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Doaa Moaz Sayem,MD, Lecturer of Anaesthesia, Department of anaesthesia, Surgical Intensive Care Unit and Pain Management Faculty of Medicine ,Beni-Suef university, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PECS block in mastectomy
Record Dates: First submitted 2022-11-10; First posted 2022-12-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Breast
Keywords: Magnesium sulphate; ketamine; PECS block; Mastectomy
MeSH Terms: conditions — Neoplasms | interventions — Mastectomy; Bupivacaine; Ketamine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Ultrasound guided pectoral nerve block will be performed after induction of general anaesthesia . Starting from the lateral third of the clavicle and moving distally and laterally to the mid axillary line. The needle will be inserted in plane with ultrasound probe between 2 pectoralis muscles and 10 mL of bupivacaine 0.25% alone or with ketamine or magnesium will be injected between the 2 pectoral after negative aspiration for blood (PECS I) then the ultrasound probe will be moved towards axilla until identification of the serratus anterior then the needle will be inserted between pectoralis minor and serratus anterior muscles and 20 mL of bupivacaine 0.25% alone or with ketamine or magnesium will be injected after negative aspiration. Skin incision will be performed 15 minutes after the block will be given . After extubation , all patients will be transferred to the post anesthesia care unit for postoperative monitoring and observation
Who Masked: Care Provider, Outcomes Assessor
Masking Description: this is a randomized double-blinded study All patients included will be divided randomly into three groups Preoperative data will be recorded by anesthesiologist who will be blinded to the study .
  The studied drugs will be prepared by anesthetist ( who will be blinded to the study and will not involved in the technique) in labeled syringes .
  Randomization will be done using a computer-generated sequence. The randomly assigned numbers in each group will be hidden in sealed and opaque envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (control group ) (Active Comparator): Patients will be given 30 mL of 0.25% bupivacaine hydrochloride in pectoral nerve block .
  Interventions: Drug: Use of Bupivacaine in pectoral nerve block in mastectomy
- Group B ( Ketamine group) (Active Comparator): Patients will be given 30 mL of 0.25% bupivacaine hydrochloride plus ketamine hydrochloride (1 mg/kg) in pectoral nerve block .
  Interventions: Drug: use of Ketamine as adjuvants to bupivacaine in pectoral nerve block in mastectomy
- Group C (Magnesium sulfate group) (Active Comparator): Patients will be given 30 mL 0.25% bupivacaine hydrochloride plus magnesium sulfate ( 28 ml bupivacaine 0.25% plus 2ml magnesium sulfate (50%) in pectoral nerve block
  Interventions: Drug: Use of Magnesium Sulfate as adjuvants to bupivacaine in pectoral nerve block in mastectomy

INTERVENTIONS:
Drug: Use of Bupivacaine in pectoral nerve block in mastectomy — Pectoral nerve block will be performed and patients will be given 30 mL of 0.25% bupivacaine hydrochloride and It will be divided into 10 mL injected between the 2 pectoral muscles on the interfascial plane, and 20 mL will be injected between the pectoralis minor and the serratus anterior muscles
  Other Names: marcain
  Arms: Group A (control group )
Drug: use of Ketamine as adjuvants to bupivacaine in pectoral nerve block in mastectomy — Pectoral nerve block will be performed and Patients will be given 30 mL of 0.25% bupivacaine hydrochloride plus ketamine hydrochloride (1 mg/kg) and It will be divided into 10 mL injected between the 2 pectoral muscles on the interfascial plane, and 20 mL will be injected between the pectoralis minor and the serratus anterior muscles
  Other Names: ketalar
  Arms: Group B ( Ketamine group)
Drug: Use of Magnesium Sulfate as adjuvants to bupivacaine in pectoral nerve block in mastectomy — Pectoral nerve block will be performed and Patients will be given 30 mL 0.25% Bupivacaine hydrochloride plus Magnesium Sulfate ( 28 ml Bupivacaine 0.25% plus 2ml magnesium sulfate 50%) and It will be divided into 10 mL injected between the 2 pectoral muscles on the interfascial plane, and 20 mL will be injected between the pectoralis minor and the serratus anterior muscles
  Other Names: Mgso4
  Arms: Group C (Magnesium sulfate group)

SUMMARY:
There are no published article that compare magnesium sulfate and ketamine as adjuvants to bupivacaine in PECS block , so the aim of this study is to evaluate the efficacy of Magnesium sulfate versus ketamine when added to local anesthetic ( Bupivacaine) in pectoral nerve block during mastectomy and detect which of these drugs has the more effective analgesic effect and decrease opioid consumption .

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in females, and its incidence increases with increase the age of the patients and it is the most expected cause of death in the world .

Surgery is the main treatment of breast cancer and other treatments include chemotherapy, radiotherapy , hormonal therapy and biological therapy or combination treatment and this depends on the type of the cancer and its stage .

Breast surgery is usually associated with significant postoperative pain. Poorly controlled postoperative pain has a negative physiological and psychological impacts as it is associated with an increase in hospital stay , medical care cost, significant postoperative nausea and vomiting , development of chronic pain syndrome and impaired quality of life .

Several methods have been involved in postoperative pain control including multi modal analgesia using multiple medication with different mechanism of action as intravenous and oral opioids , non-steroidal anti-inflammatory drugs and local anesthetic infiltration also has an important role in pain control .

Regional anesthetic procedures have an effective role in acute pain control as thoracic epidural and thoracic paravertebral block are considered the gold standard procedures for postoperative pain management for breast cancer surgery, but not every anesthesiologist is comfortable making these invasive procedures .

Recently, the pectoral nerves blocks (PECS I and PECS II) are recommended for providing intraoperative and postoperative pain control during and after breast surgery. These blocks may be more effective when compared to other regional anesthetic procedures .

Pectoral nerves blocks includes 2 types (PECS I and PECS II). The PECS block type I is a easy and reliable performed by injection an interfacial plane between the pectoralis major and pectoralis minor muscles to block the lateral region of the breast to provide analgesia for breast surgery .

The PECS block type II "modified Pecs's block'' is performed by injection at the interfascial plane between the pectoralis minor muscle and serratus anterior muscle . It aims at blocking the pectoral nerves, the intercostobrachial , intercostals (III, IV, V, and VI), and the long thoracic nerve and these are required to block the axilla also provides analgesia to mammary glands and the skin from the T2-T6 dermatomes extending into the mid-axillary line providing complete analgesia during breast surgery and several types of mastectomies .

Pectoral nerve block is usually performed using an in-line needling technique by ultrasound guidance, which is essential to identify the plane between the pectoralis major, minor muscles, and serratus anterior as well as the anatomical landmarks associated with them .

Hematoma and local anesthetic toxicity and risk of pneumothorax are adverse effects in pectoral nerve block especially PECS II block which may be reduced by using ultrasound guidance and decreasing anesthetic drug concentrations .

Various adjuvants, as fentanyl, morphine, tramadol, epinephrine, α2 agonists, dexamethasone, midazolam, neostigmine and sodium bicarbonate have been added to local anesthetics agents to prolong the time and potency of postoperative analgesia and this is may be associated with adverse effects, and the outcomes have been inadequate.

An understanding of pain mechanisms points to the role of central sensitization and N-methyl-D-aspartate (NMDA) receptor activation by excitatory amino acid transmitters in postsurgical pain .

Magnesium sulfate (MgSO4) is a non-competitive antagonist of the N-methyl-D-aspartate (NMDA) receptor in the central and peripheral nervous system, and is found to decrease the intraoperative and postoperative analgesic consumption and also it increases the duration and potency of analgesia when combined with different local anesthetics.

Magnesium augments local anesthetics (LA) action in the peripheral nerves by increasing the firing threshold in both myelinated and unmyelinated axons increasing the transmembrane potential causing hyperpolarization and adding of magnesium to bupivacaine produces an enhancement of nerve blocking .

Ketamine is also a non-competitive antagonist of the N-methyl-D-aspartate NMDA receptor antagonist commonly used for its analgesic and anesthetic effect .

Ketamine decreases the intensity of postoperative pain, reduces 24-hour opioid consumption, and delays the time to first request of analgesic therapy .

Bupivacaine is an amide local anesthetic with a slow onset, long duration of action and high potency. The maximum recommended single bolus dose of bupivacaine is 2.5 mg/Kg, bupivacaine exert its action through impairing sodium influx across the neuronal membrane by blocking the sodium channels .

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Age from 30 to 70 years old
* American Society of Anesthesiologists (ASA) I-II

Exclusion Criteria:

* Cognitive impairment
* History of alcohol or drug abuse
* Allergy to the studied drugs
* Patients with coagulation disorders
* Block site infection
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Body Mass Index( BMI) more than 30 kg/m2

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
The postoperative time to first request of analgesia | up to 24 hours
  the aim of this study is to evaluate the efficacy of Magnesium sulfate versus ketamine when added to local anesthetic (Bupivacaine) in pectoral nerve block during mastectomy and the first time of request of analgesia postoperative in hours is the primary outcome

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) , the scale is determined by measuring the distance in millimeter (mm) on the 10 centimeter (cm) line between the 0 (no pain ) and the mark of the patient . | up to 24 hours
  All patients will be followed up and assessed at baseline, one hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hours, postoperative for Visual Analogue Scale (VAS) to assess the pain intensity ,The Visual Analogue Scale VAS consists of a 10 cm line with two end points representing 0(no pain ) and 10 (worst pain )
Postoperative analgesic requirements( (pethidine in milligram/ kilogram (mg/kg) ) | up to 24 hours
  All patients will be followed up and assessed at baseline, one hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hours, postoperative for visual analogue scale to assess pain intensity and pethidine will be given 0.2-0.5 mg/kg if visual analogue scale (VAS) scale ≥ 3)
Postoperative heart rate (Beat/minute) | up to 24 hours
  All patients will be followed up and assessed at baseline, one hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hours, postoperative for heart rate measurement (Beat/minute)
Postoperative non invasive mean arterial blood pressure in millimeters of mercury (mmHg) | up to 24 hours
  All patients will be followed up and assessed at baseline, one hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hours, postoperative for non invasive blood pressure measurement in millimeters of mercury (mmHg)
Postoperative respiratory rate (breath /minute ) | Up to 24 hours
  All patients will be followed up and assessed at baseline and one hour, 2 hour, 4 hour, hour, 12 hour and 24 hours for postoperative respiratory rate measurement (breath /min)
Postoperative Nausea and Vomiting | Up to 24 hours
  All patients will be followed up and assessed at baseline, one hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hours, postoperative for postoperative Nausea and Vomiting (PONV) score (0=no nausea and vomiting, 1=mild nausea, 2=severe nausea, 3=vomiting once, and 4=repeated vomiting) .

CONTACTS AND LOCATIONS:
Overall Officials: Doaa M Khalil, lecturer, Study Director — Research Ethical Committee,faculty of medicine Beni-Suef university
Locations (1):
- faculty of medicine ,Beni-Suef university, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected Individual Participant Data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: the data will be available within 10 months
Access Criteria: individual participant data will be shared as study protocol and statistical analysis in web site
URL: http://med.bsu.edu.eg

REFERENCES:
- [Result] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- See also: Pectoral Nerves Blocks for Post-Operative Analgesia after Breast Cancer Surgery — https://mjcu.journals.ekb.eg/article_152001_92fe360f3293fe689260809014ed7a1a.pdf